CLINICAL TRIAL: NCT04999007
Title: Artificial Intelligence-assisted Decision Making for Temporary Ileostomy: A Prospective Randomized Controlled Trail.
Brief Title: Artificial Intelligence Assists Surgeons' Decision Making
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jichao Qin (Other)
Responsible Party: Sponsor-Investigator, Jichao Qin, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: TJ-IRB20210643
Record Dates: First submitted 2021-08-08; First posted 2021-08-10 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Rectal Cancer
Keywords: artificial intelligence,; rectal cancer; temporary ileostomy; anastomotic leakage
MeSH Terms: conditions — Rectal Neoplasms; Anastomotic Leak

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Whether the patients in the control arm will receive a temporary ileostomy depends on surgeons' experience.
- Intervention (Experimental): Whether the patients in the intervention arm will receive a temporary ileostomy depends on the risk of anastomotic leakage calculated by the artificial intelligence algorithm.
  Interventions: Other: Artificial intelligence algorithm

INTERVENTIONS:
Other: Artificial intelligence algorithm — Temporary ileostomy will be performed in the patients with high-risk of anastomotic leakage and not performed in the patients with low-risk of anastomotic leakage.
  Arms: Intervention

SUMMARY:
This study will evaluate whether artificial intelligence technique reduces the temporary ileostomy rate in patients with rectal cancer who receive anterior resection.

DETAILED DESCRIPTION:
Anastomotic leakage is a serious and life-threatening complication after anterior resection in patients with rectal cancer, and temporary ileostomy was introduced to reduce the serious consequences due to anastomotic leakage. However, whether a temporary ileostomy is applied in the surgery depends on the surgeon's experience, and there are no clinical guidelines to follow. Recently, artificial intelligence has widely been applied in medical field and produced some exciting results, and we have developed a high-performance artificial intelligence model based on 2369 rectal cancer patients, which showed good discrimination of anastomotic leakage and may reduce the temporary ileostomy rate. Hence, this randomized controlled trail will evaluate the artificial intelligence model for guiding surgical decision-making of performing a temporary ileostomy in patients with rectal cancer who receive anterior resection.

ELIGIBILITY:
Inclusion Criteria:

1. Aged older than 18 years and younger than 85 years.
2. Primary rectal adenocarcinoma confirmed by preoperative pathology result.
3. Expected curative resection via total mesorectal excision procedure.
4. American Society of Anesthesiologists (ASA) class I, II, or III.
5. Written informed consent.

Exclusion Criteria:

1. Pregnant or breastfeeding women.
2. Severe mental disorder or language communication disorder.
3. Hartmann surgery or colostomy is performed intraoperatively.
4. Interrupted of surgery for more than 30 minutes due to any cause.
5. Malignant tumors with other organs

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 616 (Estimated)
Dates: Start 2021-09-02 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
The rate of temporary ileostomy. | Intraoperative period
The morbidity of anastomotic leakage. | 30 days
  The diagnosis of anastomotic leakage is determined when the passage of fecal material from pelvic drainage tube or the water-soluble contrast agent enema and extra-rectal imaging. Alternatively, anastomotic leakage can be diagnosed when the integrity of the anastomosis is interrupted or the appearance of pelvic abscess next to the anastomosis by computerized tomography (CT) examination or secondary surgical exploration.

CONTACTS AND LOCATIONS:
Overall Officials: Jichao Qin, MD, Principal Investigator — Huazhong University of Science and Technology
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No